CLINICAL TRIAL: NCT02951130
Title: Milrinone in Congenital Diaphragmatic Hernia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0057; UG1HD034216 (NIH); UG1HD027904 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD027851 (NIH); UG1HD087229 (NIH); UG1HD053109 (NIH); UG1HD068278 (NIH); UG1HD068244 (NIH); UG1HD068263 (NIH); UG1HD027880 (NIH); UG1HD053089 (NIH); UG1HD087226 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2016-10-14; First posted 2016-11-01 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Congenital Diaphragmatic Hernia; Persistent Pulmonary Hypertension of the Newborn; Hypoxemic Respiratory Failure; Pulmonary Hypoplasia
Keywords: CDH; PPHN; HRF
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Persistent Fetal Circulation Syndrome; Respiratory Insufficiency | interventions — Milrinone; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Milrinone (Experimental): Milrinone infusion at 0.33µg/kg/min. The dose of the study drug will be increased to 0.66 µg/kg/min if oxygenation index (OI) remains ≥ 10 without any evidence of hypotension (as defined by the protocol) two hours after initiation of study drug. Infusion will be continued until the OI decreases to < 7. The maximum duration of study drug infusion is 72 hours.
  Interventions: Drug: Milrinone
- 5% dextrose (D5W) (Placebo Comparator): An equivalent volume of 5% dextrose (D5W) will be used for infants randomized to the placebo arm.
  Interventions: Drug: Placebo (5% Dextrose)

INTERVENTIONS:
Drug: Milrinone — The study intervention is an intravenous infusion of milrinone or placebo
  Other Names: Milrinone Lactate Injection; Primacor
  Arms: Milrinone
Drug: Placebo (5% Dextrose) — The study intervention is an intravenous infusion of milrinone or placebo
  Other Names: D5W
  Arms: 5% dextrose (D5W)

SUMMARY:
Infants with congenital diaphragmatic hernia (CDH) usually have pulmonary hypoplasia and persistent pulmonary hypertension of the newborn (PPHN) leading to hypoxemic respiratory failure (HRF). Pulmonary hypertension associated with CDH is frequently resistant to conventional pulmonary vasodilator therapy including inhaled nitric oxide (iNO). Increased pulmonary vascular resistance (PVR) can lead to right ventricular overload and dysfunction. In patients with CDH, left ventricular dysfunction, either caused by right ventricular overload or a relative underdevelopment of the left ventricle, is associated with poor prognosis. Milrinone is an intravenous inotrope and lusitrope (enhances cardiac systolic contraction and diastolic relaxation respectively) with pulmonary vasodilator properties and has been shown anecdotally to improve oxygenation in PPHN. Milrinone is commonly used during the management of CDH although no randomized trials have been performed to test its efficacy. Thirty percent of infants with CDH in the Children's Hospital Neonatal Database (CHND) and 22% of late-preterm and term infants with CDH in the Pediatrix database received milrinone. In the recently published VICI trial, 84% of patients with CDH received a vasoactive medication. In the current pilot trial, neonates with an antenatal or postnatal diagnosis of CDH will be randomized to receive milrinone or placebo to establish safety of this medication in CDH and test its efficacy in improving oxygenation.

DETAILED DESCRIPTION:
This is a pilot trial to determine if milrinone infusion in neonates ≥ 36 weeks' postmenstrual age (PMA) at birth with CDH would lead to an increase in PaO2 with a corresponding decrease in OI by itself or in conjunction with other pulmonary vasodilators such as iNO at 24 h post-infusion.

ELIGIBILITY:
Eligibility criteria:

Infants are eligible if they meet all of the following criteria:

* ≥ 36 0/7 weeks PMA by best obstetric estimate AND birth weight of ≥ 2000g
* postnatal age ≤7 days (168 hours of age)
* invasive mechanical ventilation (defined as ventilation with an endotracheal tube) and
* one arterial blood gas with an OI ≥ 10 (after tracheal tube obstruction and other easily resolvable mechanical causes for increased OI are ruled out) on the most recent arterial blood gas within 12 hours prior to the time of randomization.
* if an arterial blood gas is not available at the time of randomization, a preductal OSI of ≥ 5 can be used as an inclusion criterion instead of OI ≥ 10; (the OSI should be based on the most recent preductal pulse oximetry recording and must be within 12 hours of randomization)
* postnatal blood gas with PCO2 ≤ 80 mmHg (arterial, capillary or venous blood gas) on the most recent blood gas sample obtained within 12 hours prior to randomization Note: Criteria (iv) to (vi) must be met at the most recent analysis within 12 hours prior to randomization.

Exclusion Criteria:

Infants are ineligible if they meet any of the following criteria:

* known hypertrophic cardiomyopathy

  * Note 1: infants of diabetic mothers with asymmetric septal hypertrophy can be included as long as there is no evidence of obstruction to left ventricular outflow tract on echocardiogram,
  * Note 2: infants with other acyanotic congenital heart disease (CHD) and CDH may be included in the study and will be a predetermined subgroup for analysis)
* cyanotic CHD - transposition of great arteries (TGA), total anomalous pulmonary venous return (TAPVR), partial anomalous pulmonary venous return (PAPVR), truncus arteriosus (TA), tetralogy of Fallot (TOF), single ventricle physiology - hypoplastic left heart syndrome (HLHS), tricuspid atresia, critical pulmonic stenosis or atresia etc.,
* enrolled in conflicting clinical trials (such as a randomized controlled blinded trial of another pulmonary vasodilator therapy); Note: mothers enrolled in fetal tracheal occlusion studies such as FETO may be enrolled if permitted by investigators of the fetal tracheal occlusion study; [FETO refers to fetoscopic endoluminal tracheal occlusion and involves occlusion of fetal trachea with a balloon device at mid-gestation and subsequent removal in later gestation]
* infants with bilateral CDH

  o Note 3: infants with anterior and central defects are included in the study
* associated abnormalities of the trachea or esophagus (trachea-esophageal fistula, esophageal atresia, laryngeal web, tracheal agenesis)
* renal dysfunction (with serum creatinine > 2 mg/dL not due to maternal factors) or severe oligohydramnios associated with renal dysfunction at randomization; renal dysfunction may be secondary to renal anomalies or medical conditions such as acute tubular necrosis
* severe systemic hypotension (mean blood pressure < 35 mm Hg for at least 2 h with a vasoactive inotrope score of > 30)
* decision is made to provide comfort/ palliative care and not full treatment
* Intracranial bleed (including the following findings on the cranial ultrasound)

  * Cerebral parenchymal hemorrhage
  * Blood/echodensity in the ventricle with distension of the ventricle
  * Periventricular hemorrhagic infarction
  * Posterior fossa hemorrhage
  * Cerebellar hemorrhage
* persistent thrombocytopenia (platelet count < 80,000/mm3) despite blood product administration on the most recent blood draw prior to randomization
* coagulopathy (PT INR > 1.7) despite blood product administration on the most recent blood draw (if checked - there is no reason to check PT for the purpose of this study)
* aneuploidy associated with short life span (such as trisomy 13 or 18) will not be included in the study (infants with trisomy 21 can be included in the study)
* elevated arterial, venous or capillary PCO2 > 80 mmHg in spite of maximal ventilator support (including high frequency ventilation) on the most recent blood gas obtained within 12 hours prior to randomization
* use of milrinone infusion prior to randomization (the use of other inhaled pulmonary vasodilators such as iNO, inhaled epoprosternol, inhaled PGE1 and oral such as endothelin receptor antagonists is permitted - Note: it is unlikely to be on oral pulmonary vasodilators early in the course of CDH)
* ongoing therapy with parenteral (intravenous or subcutaneous) pulmonary vasodilators such as IV/SQ prostacyclin analogs (Epoprostenol - Flolan or Treprostinil - Remodulin or PGE1 - Alprostadil) or IV phosphodiesterase 5 inhibitors (sildenafil - Revatio) at the time of randomization. In addition, initiation of therapy with these two classes of parenteral medications during the first 24 hours of study drug initiation is not permitted and will be considered a protocol deviation. The risk of systemic hypotension is high during the first 24 hours of study-drug (milrinone) infusion and hence parenteral administration of other pulmonary vasodilators is avoided to minimize risk of hypotension.
* Subjects already on ECMO or patients who are being actively considered for ECMO by the neonatal or surgical team
* attending (neonatal, critical care or surgical) refusal for participation in the trial (including concern about presence of hemodynamic instability)

Ages: 0 Hours to 168 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satyan Lakshminrusimha, M.D., Principal Investigator — University of California, Davis
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Children's Mercy, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Per NIH Data Sharing Plan

REFERENCES:
- [Derived] Lakshminrusimha S, Keszler M, Kirpalani H, Van Meurs K, Chess P, Ambalavanan N, Yoder B, Fraga MV, Hedrick H, Lally KP, Nelin L, Cotten M, Klein J, Guilford S, Williams A, Chaudhary A, Gantz M, Gabrio J, Chowdhury D, Zaterka-Baxter K, Das A, Higgins RD. Milrinone in congenital diaphragmatic hernia - a randomized pilot trial: study protocol, review of literature and survey of current practices. Matern Health Neonatol Perinatol. 2017 Nov 27;3:27. doi: 10.1186/s40748-017-0066-9. eCollection 2017. PMID 29209510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Milrinone | 5% dextrose (D5W)
Started | 33 | 33
Completed | 32 | 32
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milrinone | 5% dextrose (D5W) | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Customized [Median (Inter-Quartile Range); unit: hours] — Age at Drug Initiation Population: Two participants did not receive any study drug.
  hours
    number analyzed (Participants) | 32 | 32 | 64
    (all) | 14.4 [9.5 to 22.2] | 19.6 [10.9 to 35.9] | 16.9 [9.9 to 27.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 16 | 20 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 29 | 23 | 52
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 30 | 25 | 55
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Oxygenation Response
Description: The primary outcome of this study is change in oxygenation from baseline (prior to study drug infusion) to 24 hours after initiation of study drug infusion. Oxygenation is assessed by oxygenation index (OI = mean airway pressure x oxygen concentration in % / PaO2 in mmHg). Oxygen saturation index (OSI = mean airway pressure x oxygen concentration in % / oxygen saturation in %) values were converted to OI values for this measure. Data are presented as OI at 24 hours minus OI at baseline. A negative value indicates improvement in oxygenation. A positive value indicates deterioration in oxygenation.
Time Frame: 24 h after initiation of study drug
Measure: Median (Inter-Quartile Range); unit: Change in Oxygenation Index
Arm/Group | Milrinone | 5% dextrose (D5W)
Number analyzed (Participants) | 32 | 32
Change in Oxygenation Index | 4.2 [-1.5 to 9] | 2.6 [0 to 9.6]

2. Secondary Outcome: Oxygenation Response at 48 and 72 h
Description: Oxygenation index at 48 and 72 h (or OI at the time of initiation of ECMO or immediately prior to death, for infants placed on ECMO or died before these time points)
Time Frame: 48 and 72 h after initiation of study drug
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Estimated Systolic Pulmonary Arterial Pressure on Echocardiogram
Description: Changes in echocardiogram to assess pulmonary arterial pressure (as defined by protocol) between pre-study drug echocardiogram and echocardiogram obtained between 24 and 72 h after starting the study drug. The outcome will be available only for those infants who have a pre-study drug echocardiogram and a second echocardiogram between 24 and 72 hours after initiation of study drug performed for clinical reasons.
Time Frame: Prior to initiation of study drug to between 24 and 72 hours after initiation of study drug
Reporting Status: Not Posted

4. Secondary Outcome: Vasoactive Inotrope Score and Systemic Blood Pressure
Description: Vasoactive Inotrope Score is a quantitative assessment of the degree of therapeutic support required by the patient to maintain adequate perfusion and/or blood pressure.
Time Frame: 72 hours after initiation of study drug
Reporting Status: Not Posted

5. Secondary Outcome: Area Under the Curve for Inspired Oxygen
Description: Area under the curve for inspired oxygen after initiation of the study drug (inspired oxygen and ventilator data from 4 time points per day - every 6 hours will be recorded to calculate area under the curve)
Time Frame: After initiation of the study drug at 4 time points per day - every 6 hours x 72 hours or discontinuation of study drug (whichever comes first)
Reporting Status: Not Posted

6. Secondary Outcome: Oxygenation Response to Additional Inotropes or Pulmonary Vasodilators
Description: If subsequent to the study drug, any additional inotrope or pulmonary vasodilator is used (such as iNO), we will evaluate the oxygenation response to these agents. If inotropes or vasodilators were used prior to the initiation of study drug, similar values will be recorded. The OI and PaO2/ FiO2 ratio prior to at least 30 min after initiation of the inotrope / vasodilator are recorded. The change in OI and PaO2/ FiO2 ratio in response to these agents is evaluated as a continuous variable and arbitrarily classified into responders, partial responders and non-responders
Time Frame: Through 24 h post study drug initiation
Reporting Status: Not Posted

7. Secondary Outcome: Supplemental Continuous Oxygen
Description: The use of supplemental oxygen at 28 d will be used to calculate the incidence of chronic lung disease. Chronic lung disease severity will be classified similar to the BPD classification in preterm infants at > 32 week gestation.
Time Frame: 28 days and 56 days postnatal age (or discharge whichever comes first)
Reporting Status: Not Posted

8. Secondary Outcome: Survival to Discharge Without ECMO
Time Frame: Measured by no ECMO at time of hospital discharge or at the time the infant reaches 120 days of life and remains in the hospital, whichever comes earlier
Reporting Status: Not Posted

9. Secondary Outcome: Clinical Status (Pulmonary and Nutritional)
Description: Clinical status - pulmonary (use of supplemental oxygen or respiratory medications - diuretics, methylxanthines, steroids, inhaled or nebulized steroids or bronchodilators) and nutritional (weight, length, head circumference, use of anti-reflux medications)
Time Frame: All clinical status measures (as defined by protocol) will be obtained just prior to the infants discharge from the hospital and again at 12 months of age.
Reporting Status: Not Posted

10. Secondary Outcome: Feasibility and Sample Size Calculation to Perform a Definitive Trial (Primary Outcome - Improvement in Survival Without ECMO
Time Frame: From initial recruitment: 16 patients enrolled per month to complete the trial in 4 years
Reporting Status: Not Posted

11. Secondary Outcome: Feasibility to Perform a Definitive Trial (Incidence of Systemic Hypotension)
Time Frame: From initial recruitment: 16 patients enrolled per month to complete the trial in 4 years
Reporting Status: Not Posted

12. Secondary Outcome: Feasibility to Perform a Definitive Trial (Incidence of Intracranial Bleeding)
Time Frame: From initial recruitment: 16 patients enrolled per month to complete the trial in 4 years
Reporting Status: Not Posted

13. Secondary Outcome: Feasibility to Perform a Definitive Trial (Incidence of Arrhythmias)
Time Frame: From initial recruitment: 16 patients enrolled per month to complete the trial in 4 years
Reporting Status: Not Posted

14. Secondary Outcome: Adjusted Oxygen Response
Time Frame: 24 h after initiation of study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study specified adverse events (AE) are monitored during the study (e.g. from treatment initiation through 24 hours after discontinuation of study drug infusion).
Arm/Group | Milrinone | 5% dextrose (D5W)
All-Cause Mortality (participants affected / at risk) | 7/33 | 2/33
Serious Adverse Events (participants affected / at risk) | 5/33 | 3/33
Other Adverse Events (participants affected / at risk) | 5/33 | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milrinone (N=33) | 5% dextrose (D5W) (N=33)
Shock (Vascular disorders) | 1 (1) | 2 (2)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milrinone (N=33) | 5% dextrose (D5W) (N=33)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 4 (4) | 1 (1)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT02951130/Prot_SAP_001.pdf
  • Informed Consent Form (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02951130/ICF_000.pdf